CLINICAL TRIAL: NCT05263934
Title: A 52-week, Randomized, Double-blind, Double-dummy, Parallel-group, Multi-centre, Non-inferiority Study to Investigate the Efficacy and Safety of Depemokimab Compared With Mepolizumab in Adults With Relapsing or Refractory Eosinophilic Granulomatosis With Polyangiitis (EGPA) Receiving Standard of Care (SoC) Therapy
Brief Title: Efficacy and Safety of Depemokimab Compared With Mepolizumab in Adults With Relapsing or Refractory Eosinophilic Granulomatosis With Polyangiitis (EGPA)
Acronym: OCEAN
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 217102; 2023-510019-20-00 (Other: EU CT Number)
Record Dates: First submitted 2022-02-28; First posted 2022-03-03 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Eosinophilic Granulomatosis With Polyangiitis
Keywords: Depemokimab; Mepolizumab; Eosinophilic Granulomatosis with Polyangiitis
MeSH Terms: conditions — Churg-Strauss Syndrome | interventions — mepolizumab

STUDY DESIGN:
Intervention Model Description: Participants will receive either depemokimab plus placebo matching mepolizumab or mepolizumab plus placebo matching depemokimab
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants receiving depemokimab+placebo matching mepolizumab (Experimental)
  Interventions: Biological: Depemokimab; Drug: Placebo matching mepolizumab
- Participants receiving mepolizumab+placebo matching depemokimab (Active Comparator)
  Interventions: Biological: Mepolizumab; Drug: Placebo matching depemokimab

INTERVENTIONS:
Biological: Depemokimab — Depemokimab will be administered
  Arms: Participants receiving depemokimab+placebo matching mepolizumab
Biological: Mepolizumab — Mepolizumab will be administered
  Arms: Participants receiving mepolizumab+placebo matching depemokimab
Drug: Placebo matching mepolizumab — Placebo matching to mepolizumab will be administered.
  Arms: Participants receiving depemokimab+placebo matching mepolizumab
Drug: Placebo matching depemokimab — Placebo matching to depemokimab will be administered.
  Arms: Participants receiving mepolizumab+placebo matching depemokimab

SUMMARY:
This study aims to investigate the efficacy and safety of depemokimab compared with mepolizumab in adults with relapsing or refractory EGPA receiving SoC therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participant (male or female) must be 18 years of age or older at the time of signing the informed consent.
* Participants who are >=40 kilogram at Screening Visit 1.
* Participants with a documented diagnosis of EGPA for at least 6 months based on the history or presence of: asthma plus eosinophilia defined as >1.0*10^9/Liter (L) and/or >10 percentage (%) of leucocytes plus at least 2 of the following additional features of EGPA: a biopsy showing histopathological evidence of eosinophilic vasculitis, or perivascular eosinophilic infiltration, or eosinophil-rich granulomatous inflammation, neuropathy, mono or poly (motor deficit or nerve conduction abnormality), pulmonary infiltrates, non-fixed, sino-nasal abnormality, cardiomyopathy (established by echocardiography or magnetic resonance imaging), glomerulonephritis (hematuria, red cell casts, proteinuria), alveolar hemorrhage (by bronchoalveolar lavage), palpable purpura, anti-neutrophil cytoplasmic antibodies positive Myeloperoxidase or Proteinase 3.
* History of relapsing OR refractory disease.
* Participants must be on a stable dose of oral prednisolone or prednisone of >=7.5 mg/day (but not >50 mg/day) or equivalent for at least 4 weeks prior to Baseline (Visit 2).
* If participants receiving immunosuppressive therapy (excluding cyclophosphamide) the dosage must be stable for the 4 weeks prior to Baseline (Visit 2) and during the study.
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies: Is a woman of non-childbearing potential (WONCBP) OR Is a woman of childbearing potential (WOCBP) and using a contraceptive method that is highly effective, with a failure rate of <1%.
* Capable of giving signed informed consent

Exclusion Criteria:

* Participants diagnosed with granulomatosis with polyangiitis; previously known as Wegener's granulomatosis or microscopic polyangiitis.
* Participants with organ-threatening EGPA as per EULAR criteria,
* Imminently life-threatening EGPA disease within 3 months prior to Screening (Visit 1).
* A current malignancy or previous history of cancer in remission for less than 12 months prior to Screening.
* Participants with alanine aminotransferase >2*upper limit of normal (ULN) or if participant is on background methotrexate or azathioprine >3*ULN, aspartate aminotransferase >2*ULN or if participant is on background methotrexate or azathioprine >3*ULN, alkaline phosphatase >=2.0*ULN, total bilirubin >1.5*ULN (isolated bilirubin >1.5*ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%), Cirrhosis or current unstable liver or biliary disease per investigator assessment.
* Participants who have severe or clinically significant cardiovascular disease uncontrolled with standard treatment.
* Participants who have known, pre-existing, clinically significant system abnormalities that are not associated with EGPA and are uncontrolled with standard treatment.
* Clinically significant abnormality in the hematological, biochemical or urinalysis screen at Visit 1.
* Chronic or ongoing active infectious disease requiring systemic treatment.
* Participants with a known, pre-existing parasitic infestation within 6 months prior to Screening Visit 1.
* A known immunodeficiency (e.g., human immunodeficiency virus [HIV]).
* Participants that, according to the investigator's medical judgment, are likely to have active coronavirus disease 2019 (COVID-19) infection. Participants with known COVID-19 positive contacts within the past 14 days must be excluded for at least 14 days following the exposure during which the participant must remain symptom-free.
* Participants with a known allergy or intolerance to a monoclonal antibody or biologic therapy or any of the excipients of the investigational products.
* Participants who have a previous documented failure with anti-Interleukin-5 /Interleukin-5 receptor therapy (e.g., mepolizumab, reslizumab, benralizumab). Participants who have received monoclonal antibodies (mAb) and who have not undergone the required washout periods, prior to Visit 1.
* Participants receiving any of the following: Oral corticosteroids: Participant requires an oral corticosteroid dose of >50 mg/day prednisolone/prednisone in the 4-week period prior to Baseline (Visit 2), Intravenous (IV), intramuscular or subcutaneous (SC) corticosteroids in the 4-week period prior to Baseline (Visit 2), Omalizumab within 130 days prior to Screening (Visit 1), Cyclophosphamide (CYC): oral CYC within 4 weeks prior to Baseline (Visit 2) and IV CYC within 3 weeks prior to Baseline (Visit 2), if their total white blood cells is >=4*10^9/L (measured using the local laboratory if necessary), Rituximab within 12 months prior to Screening (Visit 1); in addition, the Participant must have shown recovery of peripheral B-cell count to within the normal range, Tezepelumab and Dupilumab with a washout period of 5 half-lives prior to Screening Visit 1, IV or SC immunoglobulin within 6 months prior to Screening (Visit 1); For China and Japan only within 12 weeks prior to Screening (Visit 1), Interferon-alpha within 6 months prior to Screening Visit 1, Anti-tumor necrosis factor therapy within 12 weeks prior to Screening Visit 1, Anti-CD52 (alemtuzumab) within 6 months prior to Screening Visit 1.
* Participants with QT interval corrected for heart rate according to Fridericia's formula (QTcF) >=450 milliseconds (msec) or QTcF >=480 msec for participants with Bundle Branch Block in the 12-lead ECG central over-read from at Screening Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2026-09-29 (Estimated); Study Completion 2026-10-27 (Estimated)

PRIMARY OUTCOMES:
Number of participants with remission (Birmingham Vasculitis Activity Score [BVAS] =0 and a dose of oral corticosteroid [OCS] less than or equal to [<=] 4 milligram [mg] per day) | Up to Week 52
  Participants must be in remission at both Weeks 36 and 52.

SECONDARY OUTCOMES:
Number of participants in each category of accrued duration of remission | Up to Week 52
  Total accrued duration of remission is the accrued number of weeks where BVAS = 0 plus OCS dose <= 4 mg/day over the 52-week intervention period. The accrued duration was categorized into zero, >0 to <12 weeks, 12 to <24 weeks, 24 to <36 weeks or more than or equal to (>=) 36 weeks.
Number of participants with total accrued duration of remission | Up to Week 52
  Total accrued duration of remission is the accrued number of weeks where BVAS = 0 plus OCS dose <= 4 mg/day over the 52-week intervention period.
Time to first EGPA relapse | Up to Week 52
  The time to first EGPA relapse will be calculated from the date of first dose of study intervention and start date of the EGPA relapse.
Number of participants receiving in each category of mean OCS dose during the last 4 weeks of study treatment period (Weeks 49 to 52) | Weeks 49 to 52
  Number of participants receiving the mean OCS dose (categorized as 0, >0 to <=4, >4 to <=7.5 or >7.5 mg/day) will be assessed during the last 4 weeks of the study treatment period (Weeks 49 to 52).
Number of participants achieving remission (BVAS = 0 and OCS <= 4 mg/day) within the first 24 weeks with continued remission until Week 52 | Up to Week 52
Number of participants achieving remission using the European League against Rheumatism (EULAR) definition (BVAS = 0 and OCS <=7.5 mg/day) at Weeks 36 and 52 | At Weeks 36 and 52
Number of participants in each category of accrued duration of remission according to the EULAR definition of remission (BVAS = 0 plus OCS <=7.5 mg/day) over 52-week intervention period | Up to Week 52
  Total accrued duration of remission according to the EULAR definition of remission is the accrued number of weeks where BVAS = 0 plus OCS dose <=7.5 mg/day over the 52 week intervention period categorized as zero weeks; >0 to <12 weeks; 12 to <24 weeks; 24 to <36 weeks or >= 36 weeks.
Number of participants with total accrued duration of remission according to the EULAR definition of remission | Up to Week 52
  Total accrued duration of remission according to the EULAR definition of remission is the accrued number of weeks where BVAS=0 plus OCS <=7.5 mg/day over the 52-week intervention period.
Number of participants with remission (BVAS=0 and OCS <=7.5 mg/day) within the first 24 weeks with continued remission until Week 52 | Up to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (67):
- United States (9):
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Norfolk, Virginia
- Argentina (2):
  - GSK Investigational Site, La Plata
  - GSK Investigational Site, San Miguel de Tucumán
- GSK Investigational Site, Graz, Austria
- Belgium (2):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Leuven
- GSK Investigational Site, São Paulo, Brazil
- GSK Investigational Site, Toronto, Ontario, Canada
- China (8):
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Guangzhou
  - GSK Investigational Site, Hefei
  - GSK Investigational Site, Nanjing
  - GSK Investigational Site, Qingdao
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Shenzhen
  - GSK Investigational Site, Wenzhou
- France (8):
  - GSK Investigational Site, Brest
  - GSK Investigational Site, La Roche-sur-Yon
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Suresnes
  - GSK Investigational Site, Toulouse
- Germany (2):
  - GSK Investigational Site, Freiburg im Breisgau
  - GSK Investigational Site, Minden
- GSK Investigational Site, Budapest, Hungary
- GSK Investigational Site, Ramat Gan, Israel
- Italy (9):
  - GSK Investigational Site, Bari
  - GSK Investigational Site, Brescia
  - GSK Investigational Site, Florence
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Pavia
  - GSK Investigational Site, Pisa
  - GSK Investigational Site, Roma
  - GSK Investigational Site, Torrette AN
  - GSK Investigational Site, Treviso
- Japan (3):
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tokyo
- Netherlands (2):
  - GSK Investigational Site, Groningen
  - GSK Investigational Site, Leiden
- Poland (3):
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Warsaw
- Portugal (2):
  - GSK Investigational Site, Lisbon
  - GSK Investigational Site, Porto
- South Korea (2):
  - GSK Investigational Site, Gwangju
  - GSK Investigational Site, Seoul
- Spain (6):
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Pamplona
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Zaragoza
- GSK Investigational Site, Malmo, Sweden
- United Kingdom (3):
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- See also: Related Info — https://gskoceanclinicaltrial.com/?utm_source=ctgov